CLINICAL TRIAL: NCT05329675
Title: Phase II Clinical Trial of Sinphar Lipucan Capsule: the Regulation of Immune Function
Brief Title: Trial of Sinphar Lipucan Capsule to Regulate Immune Function
Acronym: TSLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB110-149-A
Record Dates: First submitted 2022-04-07; First posted 2022-04-15 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-04

CONDITIONS: Nutrition, Healthy
Keywords: Lipucan; Immune; Acute Upper Respiratory Tract Infection

STUDY DESIGN:
Intervention Model Description: Study Type : Interventional (Clinical Trial) Actual Enrollment : 108 participants Allocation: Randomized Intervention Model: Parallel Assignment, matching sex, age, and performance status Primary Purpose: Number of NK cells。
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Sham Comparator): one capsule /day
  Interventions: Dietary Supplement: Sinphar Lipucan Capsule
- Arm B (Experimental): two capsule/day
  Interventions: Dietary Supplement: Sinphar Lipucan Capsule
- Arm C (Experimental): Three capsule /day
  Interventions: Dietary Supplement: Sinphar Lipucan Capsule

INTERVENTIONS:
Dietary Supplement: Sinphar Lipucan Capsule — oral Sinphar Lipucan Capsule 1# (Arm A), 2# (Arm B), or 3# (Arm C)/day for 90 days

SUMMARY:
Trial of Sinphar Lipucan Capsule to regulate immune function

DETAILED DESCRIPTION:
The immune system is the line of defense for the health of human life entities. If the function decrease, it will reduce the body's defense to outside pathogen and easily lead to the occurrence of diseases. Immune response includes two kinds of reactions: (1) The innate immune system refers to inherited, germ-line defense mechanisms that are directed against molecular components found only in micro-organisms.. (2) The humoral immune response denotes immunologic responses that are mediated by antibodies. Health hazards have always been a trend based on health awareness. Therefore, how to use a healthy diet to promote the immune system is currently the most concerned research direction.

Because of the immunomodulatory effect of " Sinphar Lipucan Capsule " in previous animal experiments (1) Promote the secretion of Th1 type cytokine by T cells and inhibit the secretion of Th2 type cytokine; 2) Promote the secretion of IFN-γ by macrophages. 3) Promote the production of OVA antigen-specific antibodies in BALB/c female mice; 4) It can inhibit the secretion of IL-10 cytokine by antigen-specific (OVA) immune cells (that is, inhibit the secretion of Th2 cytokine), we think " Sinphar Lipucan Capsule " may be beneficial in reducing the severity and incidence of Acute Upper Respiratory Tract Infection. Therefore, human clinical trials were started to confirm its clinical effects and immunomodulatory effects.

ELIGIBILITY:
Inclusion Criteria:

- Healthy Volunteers

Exclusion Criteria:

1. Evidence of chronic cardio-pulmonary disease, immune-suppression or any chronic systemic disease or disability
2. Positive pregnancy test or currently breastfeeding
3. History of autoimmune disease
4. History of allergic rhinitis
5. History of physician diagnosed eczema
6. Known allergic reaction to Poria cocos or related species,
7. Pregnancy or currently breastfeeding.
8. History of autoimmune disease or immune disorders.
9. History of asthma.
10. History of allergic rhinitis.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 20-65 years old
Enrollment: 108 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximal CD25/69 Activation (% of NK CD25/69+ Cells) | 0 day, 30th day, and 90th day
  NK cells with evidence of CD25/69 activation were assessed on 0 day, 30th day, and 3rd month. The highest percentage found on one of these days in each participant was categorized as the the maximal CD25/69 activation

SECONDARY OUTCOMES:
Maximal Levels of IFN-α(pg/ml) | 0 day, 30th day, 90th day, 180th day and 270th day
  Interferon alpha was measured on 0 day, 30th day, and 90th day in peripheral blood mononuclear cells. The highest level on any of these days in each participant was chosen as the maximal level and used for the analysis.
Maximal Levels of IFN-γ(pg/ml) | 0 day, 30th day, 90th day, 180th day and 270th day
  IFN-γ(pg/ml) was measured on 0 day, 30th day, and 90th day in peripheral blood mononuclear cells. The highest level on any of these days in each participant was chosen as the maximal level and used for the analysis.
Maximal Levels of IgG, IgA, IgE (mg/dL) | 0 day, 30th day, 90th day, 180th day and 270th day
  IgG, IgA, IgE (mg/dL) was measured on 0 day, 30th day, and 90th day in peripheral blood mononuclear cells. The highest level on any of these days in each participant was chosen as the maximal level and used for the analysis.
Number of Upper Respiratory Infections | 0 day, 30th day, 90th day, 180th day and 270th day
  Diagnosed by professional otorhinolaryngologists or Family medicine doctors
Number of Lower Respiratory Infections | 0 day, 30th day, 90th day, 180th day and 270th day
  Diagnosed by professional otorhinolaryngologists, chest medicine doctors, or Family medicine doctors
Number of Influenza-like Illnesses | 0 day, 30th day, 90th day, 180th day and 270th day
  Diagnosed by professional otorhinolaryngologists, chest medicine doctors, or Family medicine doctors
Number of Urinary Tract Infections | 0 day, 30th day, 90th day, 180th day and 270th day
  Diagnosed by professional Genitourinary doctors, or Family medicine doctors
Number of Other Infections | Time Frame: 0 day, 30th day, 90th day, 180th day and 270th day
  Diagnosed by professional Family medicine doctors
Fatigue Severity Scale (FSS) | 0 day, 30th day, 90th day, 180th day and 270th day
  Estimated by the research nurse (Scale 9-63)

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Yuan Wu, Study Director — Asia University, Taiwan
Locations (1):
- Asia University, Taichung, Please Select, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Sharing
Supporting Information: Study Protocol
Time Frame: 4/30/2025
Access Criteria: requirement with an official application